CLINICAL TRIAL: NCT05531864
Title: The Role of Continuous Low Serratus Anterior Plane Block in Hepatocellular Carcinoma Surgery: a Randomised Clinical Trial.
Brief Title: Ultrasound-guided Continuous Low Serratus Anterior Plane Block in Hepatocellular Carcinoma Surgery
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Di (Other)
Responsible Party: Sponsor-Investigator, Liu Di, Principal Investigator, The First People's Hospital of Neijiang
Organization: The First People's Hospital of Neijiang (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JF20PJ288
Record Dates: First submitted 2022-08-25; First posted 2022-09-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Liver Neoplasms; Postoperative Analgesia; Serratus Anterior Plane Block
Keywords: serratus anterior plane block; Postoperative analgesia; liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous serratus anterior plane block (Experimental): Ultrasound-guided continuous serratus anterior plane block.
  Interventions: Procedure: Ultrasound-guided continuous low serratus anterior plane block
- Single serratus anterior plane block combined with rectus sheath nerve block (Active Comparator): Ultrasound-guided single serratus anterior plane block combined with rectus sheath nerve block.
  Interventions: Procedure: Ultrasound-guided single serratus anterior plane block

INTERVENTIONS:
Procedure: Ultrasound-guided continuous low serratus anterior plane block — Low anterior serratus plane block, move the mid-axillary line 4 and 5 intercostal puncture points are moved down and the puncture is changed to 7 and 8 intercostal.
  Arms: Continuous serratus anterior plane block
Procedure: Ultrasound-guided single serratus anterior plane block — Ultrasound-guided single anterior saw plane block was performed, and a needle was injected between the 4th and 5th costals in the midaxillary line.
  Arms: Single serratus anterior plane block combined with rectus sheath nerve block

SUMMARY:
To investigate the clinical application of ultrasound-guided continuous low serratus anterior plane block in open surgery for hepatocellular carcinoma.

DETAILED DESCRIPTION:
METHODS: Patients with hepatocellular carcinoma who attended our hospital from January 2021 to April 2023 were divided into CS group and N group according to the random number table method; CS group underwent ultrasound-guided continuous low anterior serratus plane block and N group underwent ultrasound-guided single anterior serratus plane block combined with rectus abdominis sheath block; the operation time, anesthesia time, incision length, sensory block time and sensory block maintenance time were counted and recorded. Pain score (NRS) was used to detect analgesia; alanine aminotransferase (ALT), liver function aspartate aminotransferase (AST), and prothrombin time (The time of thrombin, NRS) were measured by fluorescent quantitative PCR. （The time of thrombin (APTT), total bilirubin (TBIL) levels and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years;
2. ASAI-II;
3. BMI: 18-29 kg/m2

Exclusion Criteria:

1. Combined cardiac, cerebral, hepatic, and renal failure;
2. Comorbid psychiatric and neuromuscular disorders;
3. A history of allergy to anesthetic drugs;
4. Participation in other recent clinical or drug trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Block plane | 30 minute after the surgery begins
  The effect of anesthesia after ultrasound-guided nerve block was measured using planimetry, as well as the area being anesthetized. The chest wall between T2-T9 and ice cotton balls was used to assess the extent and extent of anesthesia block.
visual analogue scale | 24 hours after surgery
  The visual analogue scale (VAS) of the patient's pain was recorded 24 hours after operation.
visual analogue scale | 48 hours after surgery.
  The visual analogue scale (VAS) of the patient's pain was recorded 48 hours after operation.
visual analogue scale | 36 hours after surgery.
  The visual analogue scale (VAS) of the patient's pain was recorded 36 hours after operation.

SECONDARY OUTCOMES:
Patient satisfaction | 48 hours after surgery.
  The patient's satisfaction with the analgesia 2 days after surgery was recorded. The analgesic effect: 1-3 as satisfactory, 4-6 as unsatisfactory, 7-10 as ineffective
Remedial analgesic drug | 24 hours after surgery.
  Whether other analgesic drugs were added within 24 hours after operation was recorded
Intraoperative blood pressure changes | 2 hours after the beginning of surgery.
  Blood pressure changes were measured directly by radial artery puncture and recorded.
  The changes in blood pressure and heart rate before and after excision and the use of intraoperative opioids.
Intraoperative heart rate changes | 2 hours after the beginning of surgery.
  The curve of the change of the operative heart rate was recorded through the anesthesia machine.

CONTACTS AND LOCATIONS:
Overall Officials: ailing wu, Doctor, Study Director — First People's Hospital of Neijiang.
Locations (1):
- The First People's Hospital of Neijiang, Neijiang, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share this research plan with other researchers
Supporting Information: Study Protocol
Time Frame: It is expected to be shared in 2023
Access Criteria: article